CLINICAL TRIAL: NCT00965900
Title: Randomized Controlled Trial Comparing Propranolol, Endoscopic Banding Ligation, and Combined Treatment to Prevent First Variceal Hemorrhage in Patients With Liver Cirrhosis
Brief Title: Endoscopic Band Ligation (EBL) Versus Propranolol for Primary Prophylaxis of Variceal Bleeding
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Korea University (Other)
Responsible Party: Principal Investigator, Soon Ho Um, Professor, Korea University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: RCTPEBL
Record Dates: First submitted 2009-08-25; First posted 2009-08-26 (Estimated); Last update posted 2017-08-23 (Actual); Status verified 2017-08

CONDITIONS: Variceal Bleeding; Cirrhosis
Keywords: Cirrhosis; Esophagus Disorders; Varicose Veins
MeSH Terms: conditions — Fibrosis; Esophageal Diseases; Varicose Veins | interventions — Propranolol; Adrenergic beta-Antagonists

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Endoscopic band ligation (Active Comparator): Endoscopic band ligation until eradication of esophageal varices with 4 weeks interval, and then follow-up endoscopy with 3-6 months interval until 36 months after enrollment
  Interventions: Procedure: Endoscopic band ligation
- Propranolol (Active Comparator): start with 20 mg b.i.d, and adjust by 20-40 mg/d reaching reduction by 25% in HR or HR ≤55/min. After reaching target HR, then follow-up according to a preset schedule (at 1, 2, 3 months after initial treatment, then every 3 months until 36 months)
  Interventions: Drug: Propranolol
- EBL+Propranolol (Active Comparator): * EBL until eradication of esophageal varices with 4 weeks interval, and then follow-up endoscopy with 3-6 months interval until 36 months after enrollment
  * start with 20 mg of propranolol b.i.d, and adjust by 20-40 mg/d reaching reduction by 25% in HR or HR ≤55/min. After reaching target HR, then follow-up according to a preset schedule (at 1, 2, 3 months after initial treatment, then every 3 months until 36 months)
  Interventions: Procedure: EBL+Propranolol

INTERVENTIONS:
Procedure: Endoscopic band ligation — * Perform EBL within 7 days after randomization
  * Apply 1-2 band/column/session to varices in the distal 5-7 cm of the esophagus till they are eradicated (disappearance or too small to apply band) with interval of 4 weeks (at 4,8,12 weeks after initial treatment)
  * Acid suppression using proton pump inhibitor until eradicated.
  * After eradication, then follow-up endoscopy according to a preset schedule (at 1, 2, 3 months after initial treatment, then every 3-6 months until 36 months).
  Other Names: EBL
  Arms: Endoscopic band ligation
Drug: Propranolol — * start with 20 mg of propranolol b.i.d
  * Adjust by 20-40 mg/day reaching reduction by 25 percent in HR or HR less than 55/min
  * After reaching target HR, then FU according to a preset schedule (at 1, 2, 3 months after initial treatment, then every 3 months until 36 months)
  Other Names: Beta blocker
  Arms: Propranolol
Procedure: EBL+Propranolol — 1. EBL
     * Perform EBL within 7 days after randomization
     * Apply 1-2 band/column/session to varices in the distal 5-7 cm of the esophagus till they are eradicated (disappearance or too small to apply band) with interval of 4 weeks (at 4,8,12 weeks after initial treatment)
     * Acid suppression using proton pump inhibitor until eradicated.
     * After eradication, then follow-up endoscopy according to a preset schedule (at 1, 2, 3 months after initial treatment, then every 3-6 months until 36 months).
  2. Propranolol
     * start with 20 mg b.i.d
     * Adjust by 20-40 mg/day reaching reduction by 25 percent in HR or HR less than 55/min
     * After reaching target HR, then FU according to a preset schedule (at 1, 2, 3 months after initial treatment, then every 3 months until 36 months)
  Other Names: EBL+Beta blocker
  Arms: EBL+Propranolol

SUMMARY:
This study is performed to compare the efficacy and safety of EBL, propranolol, and EBL combined with propranolol in patients with medium or large varices.

DETAILED DESCRIPTION:
Current guidelines recommend prophylactic treatment with propranolol or endoscopic band ligation (EBL) to prevent variceal bleeding in patients with medium or large varices. However, it is unclear which treatment is more useful in regard to prevention of variceal bleeding as well as safety. In addition, the efficacy and safety of the combination of EBL and propranolol is not still defined. This study is performed to compare the efficacy and safety of EBL, propranolol, and EBL combined with propranolol in patients with medium or large varices.

ELIGIBILITY:
Inclusion Criteria:

* Liver cirrhosis
* Age between 18 and 70 years
* Esophageal varices with high bleeding risk: more than F2 and red color sign
* No previous history of upper gastrointestinal bleeding
* No previous history of endoscopic, radiologic, or surgical therapy for varices or ascites
* Do not take beta-blocker, ACE inhibitor, or nitrate
* Child-Pugh score <12

Exclusion Criteria:

* Patients with systolic blood pressure <100 mmHg or basal heart rate <60/min
* Portal vein thrombosis
* Uncontrolled ascites or hepatic encephalopathy
* Severe coagulation disorder: prothrombin time <40% (or INR >1.7) or platelet count <30,000/mm3
* Medium or large sized gastric or duodenal varices
* Coexisting malignancy
* Severe cardiovascular disorder, renal failure, peritonitis, sepsis
* Severe erosive esophagitis, severe esophageal stricture, active gastric or duodenal ulcer
* Contraindication to beta-blocker
* Pregnancy
* Refusal to give consent to participate in the trial

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 288 (Estimated)
Dates: Start 2006-09; Primary Completion 2019-05 (Estimated); Study Completion 2021-05 (Estimated)

PRIMARY OUTCOMES:
First esophageal variceal bleeding | 3 years after enrollment
  First esophageal variceal bleeding after enrollment

SECONDARY OUTCOMES:
Mortality; Significant esophageal variceal bleeding; Upper gastrointestinal bleeding except esophageal bleeding; Adverse events | 3 years after enrollment
  Mortality; Significant esophageal variceal bleeding; Upper gastrointestinal bleeding except esophageal bleeding; Adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Soon Ho Um, Prof, Principal Investigator — Korea University
Locations (1):
- Korea University Anam Hospital, Seoul, South Korea